CLINICAL TRIAL: NCT05865392
Title: Designing With Dissemination in Mind: Development of a Theory-based Physical Activity Intervention Using the Multiphase Optimization Strategy; Aim 1, Phase 2
Brief Title: A 12-week Field Trial of the Move Physical Activity Support Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-2183; K01HL161417 (NIH)
Record Dates: First submitted 2023-04-24; First posted 2023-05-18 (Actual); Results first posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Overweight and Obesity; Physical Inactivity
MeSH Terms: conditions — Overweight; Obesity; Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Move physical activity support program (Experimental): Participants receive the Move physical activity support program over 12 weeks.
  Interventions: Behavioral: Move physical activity support program

INTERVENTIONS:
Behavioral: Move physical activity support program — The Move program includes four intervention components: 1) 3, 60-minute group-based classes, 2) 3, 45-minute individualized support sessions, 3) access to an online fitness membership, and 4) weekly mental guided imagery sessions. Participants will be asked to build up their physical activity levels up to 150 minutes/week. They will receive an online fitness center membership during this entire 12-week program.

SUMMARY:
The objective of this study is to design and refine an activity support program for overweight or obese adults called Move. The primary outcomes are feasibility and acceptability of the Move physical activity support program.

DETAILED DESCRIPTION:
The purpose of this study is to design and refine a physical activity support program called Move, designed for adults with overweight or obesity. Participants will receive a 12-week, virtual physical activity support program called Move. Move includes four intervention components: 1) 3, 60-minute group-based classes, 2) 3, 45-minute individualized support sessions, 3) access to an online fitness membership, and 4) mental guided imagery sessions. Participants will be asked to build their physical activity levels up to 150 minutes/week. The primary outcome is to evaluate the program's acceptability and feasibility from both the participant and the provider perspectives.

ELIGIBILITY:
Inclusion Criteria:

For both participant partners and the provider partner:

* Have access to a computer and/or smart phone, and Wi-Fi
* Speak English

For the participant partners only:

* Body Mass Index 25-45 kg/m2
* Insufficiently active (defined as <150 min/week of voluntary exercise at moderate intensity over the past 3 months)
* Willing not to enroll in any other formal weight loss, physical activity program, or fitness center membership over the next 5 months.
* Have a primary care physician (or has access to a healthcare professional and/or are willing to establish care with a primary care physician prior to study enrollment) to address medical issues which may arise during screening or study procedures/interventions.
* Capable and willing to give informed consent, understand exclusion criteria, attend the Move+ program sessions, and complete outcome measures.

For the provider partners only:

* >1 year experience with delivering lifestyle interventions involving changes in diet and/or exercise behaviors.

Exclusion Criteria:

For participant partners:

* Considered high risk, based on the American College of Sports Medicine Guidelines for Exercise Testing and Prescription60 (i.e. have CVD symptoms or known CVD, diabetes, or end-stage renal disease).
* Females who are currently pregnant or lactating, were pregnant within the past 3 months, or planning to become pregnant in the next 5 months will also be excluded
* Self-reported cardiovascular disease:
* Cardiac, peripheral vascular, or cerebrovascular disease
* Self-reported symptoms suggestive of cardiovascular disease:
* pain, discomfort in the chest, neck, jaw, arms, or other areas that may result from cardiac ischemia; shortness of breath at rest or with mild exertion; dizziness or syncope; orthopnea or paroxysmal nocturnal dyspnea; ankle edema; palpitations or tachycardia; intermittent claudication.
* Self-reported end-stage renal disease
* Self-reported diabetes (history of type 1 or type 2 diabetes)
* Uncontrolled hypertension, defined as diastolic blood pressure >100 mmHG, systolic blood pressure >160 mmHG, or resting heart rate >100 bpm as measured in duplicate at the screening visit after 5 minutes of rest in a seated position.
* Self-reported pulmonary disease requiring chronic oxygen supplementation; severe asthma or chronic obstructive pulmonary disease requiring hospitalization in past year.
* Plans to relocate in the next 4 months
* Currently participating in or planning to participate in any formal weight loss, dietary modification, or physical activity/exercise programs or clinical trials.
* Current severe depression or history of severe depression within the previous year, based on DSM-IV-TR criteria for Major Depressive Episode. Score > 18 on BDI will require further assessment by the Study MD to determine if it is appropriate for the subject to participate in the study.
* History of other significant psychiatric illness (e.g., psychosis, schizophrenia, mania, bipolar disorder) which in the opinion of the Study MD would interfere with ability to adhere to the exercise intervention.
* History of clinically diagnosed eating disorders including anorexia nervosa, bulimia, binge eating disorder. Score >20 on the EATS-26 or pattern of response on the QEWP-5 suggestive of possible binge eating disorder or bulimia will require further assessment by the Study MD to determine if it is appropriate for the subject to participate in the study.
* Current alcohol or substance abuse
* Nicotine use (current or past 6 months)
* Regular use of prescription or over-the-counter medications known to significantly impact appetite, weight, sleep, or energy metabolism (e.g., appetite suppressants, lithium, stimulants, anti-psychotics, tricyclic antidepressants)
* Regular use of obesity pharmacotherapeutic agents within the last 6 months.
* Previous obesity treatment with surgery or weight loss device, except: (1) liposuction and/or abdominoplasty if performed > 1 year before screening, (2) lap banding if the band has been removed > 1 year before screening, (3) intragastric balloon if the balloon has been removed > 1 year before screening (4) duodenal-jejunal bypass sleeve, if the sleeve has been removed > 1 year before screening or 5) AspireAssist or other endoscopically placed weight loss device if the device has been removed > 1 year before screening.

For provider partners:

* None

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2023-02-16 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Ostendorf, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Community Members: Participants receive the Move physical activity support program over 12 weeks.
  Move physical activity support program: The Move program includes four intervention components: 1) 3, 60-minute group-based classes, 2) 3, 45-minute individualized support sessions, 3) access to an online fitness membership, and 4) weekly mental guided imagery sessions. Participants will be asked to build up their physical activity levels up to 150 minutes/week. They will receive an online fitness center membership during this entire 12-week program.
- Coaches: Coach delivered the Move physical activity support program
Period: Overall Study
Arm/Group | Community Members | Coaches
Started | 17 | 1
Completed | 9 | 1
Not Completed | 8 | 0
Not completed — Withdrawal by Subject | 4 | 0
Not completed — Didn't meet inclusion criteria | 4 | 0

BASELINE CHARACTERISTICS:
Population: Results are only reported at the level of the community member (n=9) and not at the level of the coach (n=1) to maintain confidentiality for the coach.
Arm/Group | Community Members
Number analyzed (Participants) | 9
Age, Continuous [Mean (Full Range); unit: years] | 45.3 [35.7 to 61.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 5
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 9
Weight [Mean (Standard Deviation); unit: kg] | 89.9 (12.5)
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 33.3 (4.4)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 121.5 (12.4)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 78.5 (10.1)

OUTCOME MEASURES:

1. Primary Outcome: Acceptability of Move Program Components, Measured With the Acceptability of Intervention Measure (AIM)
Description: Scores from the Acceptability of Intervention Measure (AIM) range from 1 to 5, with higher scores indicating higher acceptability.
Time Frame: 12 weeks
Population: All participants who started the intervention (n=9 community members, n=1 coach) were included in the analysis. Since there is only 1 coach, 95% CIs are not reported at the coach level.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Coach: A coach delivered the Move physical activity support program.
Arm/Group | Community Members | Coach
Number analyzed (Participants) | 9 | 1
score on a scale
  Group-based classes | 4.14 [3.66 to 4.62] | 5
  1:1 support sessions | 4.28 [3.70 to 4.86] | 5
  Guided imagery sessions | 3.25 [2.22 to 4.28] | 4
  Online fitness membership | 4.44 [3.61 to 5.28] | 5

2. Primary Outcome: Feasibility of Move Program Components, Measured With the Feasibility of Intervention Measure (FIM)
Description: Scores from the Feasibility of Intervention Measure (AIM) range from 1 to 5, with higher scores indicating higher acceptability.
Time Frame: 12 weeks
Population: All participants who started the intervention (n=9 community members, n=1 coach) were included in the analysis. Since there is only 1 coach, 95% CIs are not reported for the coach level data.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Community Member: Participants receive the Move physical activity support program over 12 weeks.
  Move physical activity support program: The Move program includes four intervention components: 1) 3, 60-minute group-based classes, 2) 3, 45-minute individualized support sessions, 3) access to an online fitness membership, and 4) weekly mental guided imagery sessions. Participants will be asked to build up their physical activity levels up to 150 minutes/week. They will receive an online fitness center membership during this entire 12-week program.
Arm/Group | Community Member | Coach
Number analyzed (Participants) | 9 | 1
score on a scale
  Group-based classes | 4.00 [3.60 to 4.40] | 5
  1:1 support sessions | 4.08 [3.61 to 4.55] | 4.25
  Guided imagery sessions | 3.81 [2.82 to 4.79] | 4
  Online fitness membership | 4.03 [2.73 to 5.32] | 1.25

3. Primary Outcome: Acceptability of the Move Physical Activity Support Program, Measured With the Net Promoter Score (NPS)
Description: Acceptability of the Move physical activity support program will be assessed using the Net Promoter Score (NPS) from the participant and provider perspectives. The score is calculated as a composite score from responders. Each responder rates the program between 0 and 10. Each responder is categorized as promotors (scores 9-10), passives (scores 7-8), or detractors (scores 0-6). The NPS is then calculated by the [% of promoters (scores 9 or 10) minus % detractors (scores 6 or lower)] multiplied by 100. Possible scores ranges from -100 to +100. Scores >0 indicate the component is acceptable. Negative scores indicate that a higher percentage of respondents were classified as detractors (scores 6 or lower) compared to promoters (scores 9 or 10). Only one score is calculated per support program type. There is no measure of central tendency for this outcome. See https://www.netpromoter.com/know/ for more information in how this score is calculated.
Time Frame: 12 weeks
Population: All participants who started the intervention (n=9 community members, n=1 coach) were included in the analysis.
Measure: Number; unit: units on a scale
Arm/Group | Community Member | Coach
Number analyzed (Participants) | 9 | 1
units on a scale
  Group-based Class Component | 11 | 100
  1:1 support sessions | 22 | 100
  Guided imagery sessions | -22 | 0
  Online fitness membership | 56 | 0

4. Primary Outcome: Feasibility of the Move Physical Activity Support Program - Quantitative
Description: Feasibility of the Move physical activity support program will be assessed using the Perceived Characteristics of Intervention Scale (PCIS) collected only at the level of the provider. Scores range from 0 to 4, with higher scores indicating a better outcome.
Time Frame: 12 weeks
Population: The coach who delivered the Move program completed this questionnaire at 12 weeks and was included in the analysis. Community members were not asked to complete this survey. The survey was only collected at the coach level.
Measure: Number; unit: score on a scale
Arm/Group | Coach
Number analyzed (Participants) | 1
score on a scale | 3.5

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Adverse events were recorded as they occurred throughout the 12-week intervention period. Adverse event data were not collected from coaches. Adverse event data were only collected at the community member level.
Arm/Group | Community Members
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

LIMITATIONS AND CAVEATS:
As this was a pilot feasibility study, only a small number of participants were included and analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-29): https://cdn.clinicaltrials.gov/large-docs/92/NCT05865392/Prot_SAP_000.pdf